CLINICAL TRIAL: NCT05262192
Title: Assessment of Irisin Level in Cancer Anorexia Cachexia Syndrome and Improving Quality of Life With Nutrition Education
Brief Title: Nutrition Education and Quality of Life in Cancer Cachexia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, diler us altay, Assoc. Prof., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ordu55
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Cancer Cachexia
Keywords: Cancer Anorexia Cachexia Syndrome; irisin; cachectic factors
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Nutrition education will be given to the experimental group. No intervention will be applied to the control group.
Who Masked: Participant
Masking Description: Participants will not know which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Nutrition education will be given to the experimental group.
  Interventions: Other: nutrition education
- control group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: nutrition education — Nutrition education will be given to the patients in the experimental group.
  Arms: study group

SUMMARY:
With the project the investigators propose, the investigators aim to find answers to the following questions: Are some cachectic factors and cytokines associated with plasma level irisin in patients with advanced stage cancer diagnosed with CACS? Could irisin be a new cachectic factor for patients with CACS? Can providing nutritional education to these patients slow cachexia and can a quality survival be achieved in line with the data obtained from the assessment of quality of life? and the experimental approaches to find answers to these questions make this project unique.

DETAILED DESCRIPTION:
Cancer is the uncontrolled growth of a group of cells in the body. Side effects related to cancer and treatments are one of the most difficult issues for patients and physicians. Cachexia is the second cause of cancer-related deaths after sepsis. Cachexia is a condition that progresses with weight loss in cancer patients and cannot be reversed with normal nutrition. In recent years, it has been found that cancer cachexia is associated with anorexia and has been named as cancer anorexia cachexia syndrome (CACS). Along with involuntary weight loss, appetite loss is observed in CACS patients and this decreases the quality of life. CACS is most common in people with advanced disease and the occurrence of the syndrome depends on the types of cancer. Weight loss is seen before starting treatment in 50-85% of gastrointestinal, pancreatic, lung and colorectal cancers. CACS is held responsible for 20% of cancer-related deaths. Despite these conditions, it is still considered unimportant and often incurable.

The occurrence of CACS depends on many factors. It has not been fully clarified yet which biochemical mechanisms arise. In this process, cachectic factors released from tumor cells and causing muscle and fat atrophy are proteolysis inducing factor (PIF), Zinc-α-2 Glycoprotein (ZAG) and the proinflammatory cytokines (tumor necrosis factor-α (TNF-α), Interleukin-1 (IL-1), interleukin-6 (IL-6)), which are over-synthesized by the body, importance is known. However, the search for new and more precise agents to cause cachexia is still ongoing. Irisin, which causes weight loss, a newly discovered adipomyokine known to have antiinflammatory, antidiabetic, and antiobesity effects.

With the project the investigators propose, the investigators aim to find answers to the following questions: Are some cachectic factors and cytokines associated with plasma level irisin in patients with advanced stage cancer diagnosed with CACS? Could irisin be a new cachectic factor for patients with CACS? Can providing nutritional education to these patients slow cachexia and can a quality survival be achieved in line with the data obtained from the assessment of quality of life? and the experimental approaches to find answers to these questions make this project unique.

Within the scope of this project, firstly, irisin will be measured in plasma samples taken from 80 patients diagnosed with advanced cancer, who have been diagnosed with CACS together with some cachectic factors and cytokines. Randomly selected nutrition education to be given and not given patients, measurements of all determined parameters at plasma levels will be made again at specified time intervals (starting 12th week and 24th week). In addition, all patients during this process body weight, oral intake status, amount of food consumed in the last 24 hours, presence of nausea / vomiting, chewing and swallowing functions, body mass index (BMI-kg / m2), lean mass index (BMI-kg / m2), weight loss and comprehension performance status (CPS), routine biochemical tests and quality of life assessment scales will be done

If our hypothesis is realized, possible biomarker specific to CACS has been identified,nutritional education will be answered for the first time within the scope of this project to slow down CACS and provide better quality of survival during the disease. In line with the data obtained from this project, in future projects, cachectic cancer model can be created for animals, irisin injection can slow down atrophy and cachexia, and thus, quality survival can be achieved in cancer types with high attenuation. With this work, the investigatorscreate fear in the society,affect people negatively,dragging people to the bottom with the attenuation,the investigators aim to improve the life expectancy of cancer patients, that is, to increase the quality of survival.

ELIGIBILITY:
Inclusion Criteria:

* It is planned to be applied to patients with malignancy, being 18 older and including groups of similar age, clinically approved (anorexia-cachexia-clinically approved).

Exclusion Criteria:

* Patients under the age of 18, having undergone any surgical procedure in the last 4 weeks, received radiotherapy or chemotherapy treatment, received drug therapy that modulates metabolism or weight deeply, patients with different cancer diagnoses, who were followed up and treated in the outpatient clinic before, will not be included in the study group. ..

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
SF-36 Quality of Life Scale | 12 weeks
  The SF-36 Short Form was developed and made available by Rand Corporation to assess the quality of life. It was translated into Turkish in our country and its validity and reliability study was carried out by Koçyiğit et al. In addition to being short and easy to apply, the scale has a wide range of uses. SF-36 short form is frequently used to determine the quality of life in cancer patients. The SF-36 quality of life scale consists of 36 questions and eight sub-dimensions. SF-36 has 8 sub-dimensions as general health perception, physical function, physical role, pain, vitality, social function, mental role, and mental function, and 2 summary areas as mental health and physical health.
  The summary scores obtained were expressed as a continuous variable ranging from zero to one hundred. Zero indicates ill health, 100 indicates well-being. The purpose of obtaining summary scores is to facilitate interpretation and comparisons
Determination of biochemical parameters by ELISA method | 12 weeks
  After reaching a sufficient number of patients, slimming myokines, cachectic factors, and cytokines will be measured by the commercial kits ELISA (Enzyme-Linked Immunosorbent Assay) method. ELISA technique is the gold standard for quantitation of soluble proteins and provides rapid and consistent results that are easy to analyze.
Hemoglobin measurument in plasma samples | 12 weeks
  Hemoglobin (Hgb( g/dL); grams of hemoglobin per deciliter.
Body Mass Index Measurument | 12 weeks
  Especially body mass indexes of all patients weight and height will be combined to report BMI in kg/m^2 will be measured again at the beginning of the study and after the nutrition and psychological training.
C-reactive protein measurument in plasma samples | 12 weeks
  C-reactive protein (CRP(mg/L) miligrams of CRP per liter.It is possible to say that high CRP levels indicate an acute inflammatory reaction or an infection in the body, and a decrease in CRP levels indicates that the inflammatory reaction or infection has started to decrease.
Alanine transaminase measurument in plasma samples | 12 weeks
  Alanine transaminase (ALT (U/L) units of ALT per liter. Plasma ALT level is commonly measured clinically as a biomarker for liver health. The test is part of blood panels.
Aspartate transaminase measurument in plasma samples | 12 weeks
  Aspartate transaminase (AST(U/L) units of AST per liter.Plasma AST (aspartate transaminase) level is commonly measured clinically as a biomarker for liver health. The test is part of blood panels.
Urea measurument in plasma samples | 12 weeks
  Urea (mg/dL)milligrams of urea per deciliter. Blood urea nitrogen (BUN) is a medical test that measures the amount of urea nitrogen found in the blood. The liver produces urea in the urea cycle as a waste product of the digestion of protein. Normal human adult blood should contain 6 to 20 mg/dL (2.1 to 7.1 mmol/L) of urea nitrogen.
Creatinine measurument in plasma samples | 12 WEEKS
  Creatinine(mg/dL) milligrams of creatinine per deciliter. Normal creatinine values average 0.6-1.3 mg/dL. If this value is above 2.0, renal failure is considered. However, in some cases, it has been observed that the creatinine value increases due to the rapid muscle metabolism in athletes who do heavy sports.
Prealbumin measurument in plasma samples | 12 weeks
  Prealbumin(mg/dL); milligrams of prealbumin per deciliter. It is used to evaluate nutritional status. Measurement of blood prealbumin level is especially important in premature infants or people with suspected malnutrition.
Transferrin measurument in plasma samples | 12 weeks
  Transferrin(mg/dL); milligrams of transferrin per deciliter. Transferrins are glycoproteins found in vertebrates that bind to and consequently mediate the transport of iron (Fe) through blood plasma. They are produced in the liver and contain binding sites for two Fe3+ ions. The transferrin test is a laboratory test that provides information about the saturation of transferrin with iron. The transferrin test is usually ordered when iron deficiency is suspected.
albumin measurument in plasma samples | 12 weeks
  Albumin (g/dL)grams of albumin per deciliter. It is the most important protein in the blood plasma that regulates the oncotic pressure that allows large protein molecules to pass through narrow areas such as capillaries.
fibrinogen measurument in plasma samples | 12 WEEKS
  fibrinogen (mg/dL) milligrams of fibrinogen per deciliter. Fibrinogen (factor I) is a glycoprotein complex, produced in the liver, that circulates in the blood of all vertebrates.During tissue and vascular injury, it is converted enzymatically by thrombin to fibrin and then to a fibrin-based blood clot.
Ceruloplasmin measurement in plasma samples | 12 weeks
  Ceruloplasmin (mg/dL) milligrams of ceruloplasmin per deciliter. Ceruloplasmin(or caeruloplasmin) is a ferroxidase enzyme that in humans is encoded by the CP gene. Ceruloplasmin is the major copper-carrying protein in the blood, and in addition, plays a role in iron metabolism.
Alpha-1 antitrypsin measurement in plasma samples | 12 weeks
  Alpha-1 antitrypsin (mg/dL) ; milligrams of alpha-1 antitrypsin per deciliter. Alpha-1 antitrypsin deficiency (A1AD or AATD) is a genetic disorder that may result in lung disease or liver disease. The onset of lung problems is typically between 20 and 50 years of age.[This may result in shortness of breath, wheezing, or an increased risk of lung infections. Complications may include chronic obstructive pulmonary disease (COPD), cirrhosis, neonatal jaundice, or panniculitis.
Cancer antigen 15-3 measurement in plasma samples | 12 weeks
  Cancer antigen 15-3 (CA15-3) (U/mL) units of CA 15-3 per mililiter. Cancer antigen 15-3 is a protein made by a variety of cells, particularly breast cancer cells. The protein moves into the blood, where it can be measured.CA15-3 levels are higher than normal in most women with breast cancer that has spread to other parts of the body (called metastatic breast cancer). Not all types of breast cancer will cause CA 15-3 levels to rise, as some types of cancer cells don't over-produce the antigen.
Cancer antigen 19-9 measurement in plasma samples | 12 weeks
  Cancer antigen 19-9 (U/mL) units of CA 19-9 per milliliter. This test measures the amount of a protein called CA 19-9 (cancer antigen 19-9) in the blood. CA 19-9 is a type of tumor marker. Tumor markers are substances made by cancer cells or by normal cells in response to cancer in the body.
carcinoembryonic antigen (CEA) measurement in plasma samples | 12 weeks
  carcinoembryonic antigen (CEA)(ng/mL) nanograms of carcinoembryonic antigen per mililiter. Carcinoembryonic antigen (CEA) is a protein normally found in very low levels in the blood of adults. The CEA blood level may be increased in certain types of cancer and non-cancerous (benign) conditions. A CEA test is most commonly used for colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Diler US ALTAY, Assoc. Prof., Principal Investigator — Ordu University

IPD SHARING:
Plan to Share IPD: No